CLINICAL TRIAL: NCT00589654
Title: Menstrual Cycle Maintenance and Quality of Life: A Prospective Study
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 97-127; DAMD17966292
Record Dates: First submitted 2007-12-26; First posted 2008-01-10 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Amenorrhea; Menstrual Cycle; Breast Cancer
Keywords: amenorrhea; menstrual cycle; Breast cancer; questionnaire; 97-127
MeSH Terms: conditions — Amenorrhea; Breast Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Data collection instruments will be obtained at baseline and every six months. Follow-up will range between 26-42 months for participants.

SUMMARY:
Very little is known about the incidence, onset, time course, and symptomatology of premature menopause induced by breast cancer therapy. No prospective study exists. The purpose of the present study is to identify determinants of treatment-related amenorrhea nad its effect on quality of life in a cohort of youg breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Non-institutional (community dwelling) woman of any race
* Between 18-45 years at the first screening visit
* Have regular menstrual cycles
* Diagnosed with invasive breast cancer stage I, II, III within the previous eight months
* Have physician agreement for patient participation

Exclusion Criteria:

* No menstrual bleeding cycles
* Psychiatric or psychologic abnormality precluding the informed consent process or which would decrease compliance
* Previous malignancy (excepting basal and squamous skin cancer and stage 0 cervical cancer)
* Stage IV breast malignancy
* Residency outside United States
* No telephone

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Stage 1-3 breast cancer patients 18-45 years of age will be identified. Those with normal menstrual cycles will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 810 (Estimated)
Dates: Start 1997-12; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The overall goal of the proposed research is to recruit and follow young breast cancer patients aged 45 and younger, in order to examine menstrual cycle maintenance. | Conclusion of the study

SECONDARY OUTCOMES:
Examine possible predictors of treatment-related amenorrhea including age, smoking history, race, and treatment variables | Conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Tracy-Ann Moo, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org